CLINICAL TRIAL: NCT06885476
Title: Infusion of Alloreactive nk Cells for Acute Myeloid Leukemia Patients, Eligible for Allogeneic Stem Cell Transplantiation, With Persistent Minimal Residual Disease After Conventional Chemotherapy
Brief Title: Infusion of Alloreactive nk Cells for Mrd-positive Aml Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRD-NK
Record Dates: First submitted 2021-01-22; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-04

CONDITIONS: Acute Myeloid Leukemia; Minimal Residual Disease; Natural Killer Cell
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infusion of alloreactive NK cells (Experimental): Infusion of alloreactive NK cells for acute leukemia patients, eligible for allogeneic stem cell transplantation, with persistent minimal residual disease after conventional chemotherapy
  Interventions: Biological: Infusion of alloreactive NK cells

INTERVENTIONS:
Biological: Infusion of alloreactive NK cells — Infusion of alloreactive NK cells for acute leukemia patients harboring minimal residual disease after conventional chemotherapy and prior to allogeneic stem cell transplantation

SUMMARY:
This is a interventional, transplantation study. The procedure under study is the infusion of alloreactive NK cells in adult AML patients, eligible for ASCT, who achieved CR after conventional chemotherapy, but harbor MRD-positivity.

Haploidentical KIR-L mismatched donors will be included if present at least one allele mismatch at a class I locus among the following ones: HLA-C alleles with Asn77-Lys80, HLA-C alleles with Ser77-Asn80, HLA-Bw4 alleles. KIR-L mismatched donor alloreactive NK cell repertoire will be evaluated in order to determine the functional cell dose to be used for NK cell collection. Phenotypical analysis of KIRs will be correlated to functional tests. NK cells will be selected from a steady-state large volume leukapheresis product from a suitable haploidentical KIR-ligand incompatible donor. NK cell purification will be performed if the donor leukapheresis product contains at least 10x106 NK cells/Kg.

Immunomagnetic enrichment of NK cells will follow two subsequent steps: 1) depletion of CD3+ T cells followed by 2) positive selection of CD56+ NK cells.

Patients will receive immunosuppressive chemotherapy, fludarabine (Flu) 25 mg/mq/ from day -5 to -3 and cyclophosphamide (Cy) 2 g/mq on day -2 (Flu/Cy). Two days after Cy administration, patients will be infused intravenously with a single dose of cryopreserved NK cells (day 0), which will be followed by subcutaneous administration of IL-2 (10 x 106 IU/day, 3 times weekly) for 2 weeks (6 doses total). PB samples will also be collected for biological studies. In particular, PB samples will be collected for molecular assessment of microchimerism and tracking of haploidentical NK cells for 30 days, immunophenotype studies, alloreactive NK cells cloning and functional assays (cytotoxicity). Enrolled patients will be followed up for at least 12 months after NK cell infusion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of de novo or secondary AML
* Age ≥ 18 years
* Morphologic CR
* Eligibility for ASCT
* MRD-positivity after induction chemotherapy
* Availability of a KIR-L incompatible haploidentical donor
* Performance Status ≥ 70% (Karnofsky score) or ≤ 2 (WHO).
* Adequate renal (serum creatinine < 2 mg/dl), pulmonary (Sat O2 ≥ 96%) and hepatic (ALT/AST < 2.5 x N) function.
* Left Ventricular Ejection Fraction (LVEF) of >50% as determined by Echocardiogram (ECHO).
* Signed informed consent.

Exclusion Criteria:

* Diagnosis of AML FAB M3
* HIV positivity.
* HCV positivity with high viral load.
* Pregnant or nursing females.
* Current uncontrolled infection.
* Signs or symptoms of fluid retention (e.g. pleural effusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety of infusing a functional target cell dose of 2x105 alloreactive NK cells/kg in AML patients,eligible for ASCT, with persistent MRD after conventional chemotherapy | 48 months
  Safety of infusing a functional target cell dose of 2x105 alloreactive NK cells/kg in AML patients,eligible for ASCT, with persistent MRD after conventional (number of adverse events and severe adverse events)
Feasibility of collecting a functional target cell dose of 2x105 alloreactive NK cells/kg in at least 70% of patients entering the study | 48 months
  Feasibility of collecting a functional target cell dose of 2x105 alloreactive NK cells/kg in at least 70% of patients entering the study as evaluated by in vitro cytotoxicity assay.

SECONDARY OUTCOMES:
Number of patients who achieve and maintain MRD negativity after infusion of alloreactive NK cells | 48 months
  Number of patients who achieve and maintain MRD negativity after infusion of alloreactive
Number of patients who enter ASCT in MRD-negativity | 48 months
  Number of patients who enter ASCT in MRD-negativity
Relapse-free survival (RFS) of patients infused with alloreactive NK cells | 48 months
  Relapse-free survival (RFS)of patients infused with alloreactive NK cells
overall survival (OS) of patients infused with alloreactive NK cells | 48 months
  overall survival (OS) of patients infused with alloreactive NK cells
Assess the predictive impact of donor NK cell repertoire on overall survival | 48 months
  Assess the predictive impact of donor NK cell repertoire as evaluated as the number of alloreactive NK cells/kg, in terms of overall survival
Assess the predictive impact of donor NK cell repertoire on relapse-free survival | 48 months
  Assess the predictive impact of donor NK cell repertoire as evaluated as the number of alloreactive NK cells/kg, in terms of relapse-free survival
Evaluate the microchimerism of patients receiving human NK cells | 48 months
  Evaluate the microchimerism of patients receiving human NK cells, as evaluated as percent of donor's cells into recipients
Functionally evaluate, in vitro and ex vivo, the antitumor activity of infused NK cells | 48 months
  Functionally evaluate, in vitro and ex vivo, the antitumor activity of infused NK cells, as evaluated by in vitro cytotoxicity assay (percent of lysis by donor NK cells of recipients cells).
Assess the molecular features of infused NK cells | 48 months
  Assess the molecular features of infused NK cells, qualitative gene expression profile.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Curti, Principal Investigator — Istituto di Ematologia Seràgnoli, Azienda Ospedaliero-Universitaria di Bologna (IRCCS)
Locations (1):
- Antonio Curti, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No